CLINICAL TRIAL: NCT04928976
Title: A Study to Evaluate the Ability of Speech- and Language-based Digital Biomarkers to Detect and Characterise Prodromal and Preclinical Alzheimer's Disease in a Clinical Setting
Brief Title: Amyloid Prediction in Early Stage Alzheimer's Disease Through Speech Phenotyping
Acronym: AMYPRED-US
Status: Completed | Type: Observational
Sponsor: Novoic Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: NOV-0110
Record Dates: First submitted 2021-05-20; First posted 2021-06-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-06

CONDITIONS: Alzheimer Disease; Preclinical Alzheimer's Disease; Prodromal Alzheimer's Disease; Alzheimer's Disease (Incl Subtypes); Mild Cognitive Impairment
Keywords: Alzheimer's disease; Preclinical Alzheimer's disease; Prodromal Alzheimer's disease; Mild Cognitive Impairment; Normal Cognition; Amyloid; Speech; Acoustic; Language; Linguistic; Machine Learning; Artificial Intelligence
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Speech; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Arm 1: MCI amyloid positive: * Meet the National Institute of Aging - Alzheimer's Association (NIA-AA) core clinical criteria (2011) for MCI due to Alzheimer's
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 2: MCI amyloid negative: * Non-AD Mild Cognitive Impairment (MCI)
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 23-30 (inclusive)
- Arm 3: CN amyloid positive: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Positive amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)
- Arm 4: CN amyloid negative: * Absence of a diagnosis of cognitive disorder and/or subjectively reported cognitive decline
  * Negative amyloid PET or amyloid CSF status.
  * MMSE 26-30 (inclusive)

SUMMARY:
The primary objective of the study is to evaluate whether a set of algorithms analysing acoustic and linguistic patterns of speech can detect amyloid-specific cognitive impairment in early stage Alzheimer's disease, as measured by the AUC of the receiver operating characteristic (ROC) curve of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) Arms. Secondary objectives include (1) evaluating whether similar algorithms can detect amyloid-specific cognitive impairment in the cognitively normal (CN) and MCI Arms respectively, as measured on binary classifier performance; (2) whether they can detect MCI, as measured on binary classifier performance (AUC, sensitivity, specificity, Cohen's kappa), and the agreement between the PACC5 composite and the corresponding regression model predicting it in all Arms pooled (Wilcoxon signed-rank test, CIA); (3) evaluating variables that can impact performance of such algorithms of covariates from the speaker (age, gender, education level) and environment (measures of acoustic quality).

ELIGIBILITY:
Inclusion Criteria:

* Amyloid status must be known, based on an amyloid PET scan or CSF amyloid test, no older than 30 months at the time of consent for Arm 2 and Arm 4 participants (amyloid negative Arms).
* Amyloid status must be known, based on an amyloid PET scan or CSF amyloid test, no older than 60 months at the time of consent for Arm 1 and Arm 3 (amyloid positive Arms).
* Subjects must be aged 50-85 (inclusive).
* Subjects must have MMSE scores of 23-30 (inclusive) based on a test not older than 1 month at the time of the visit.
* Date of diagnosis (if applicable) maximum of five years prior to consent.
* Subjects' first language must be English.
* Willing to participate in a study investigating speech and dementia.
* Availability of a person ('caregiver') who in the investigator's judgment has frequent and sufficient in-person contact with the participant, and is able to provide accurate information regarding the participant's cognitive and functional abilities. This is most likely met when living with a caregiver.
* Able to provide valid informed consent.
* Able to use, or has a caregiver who is able to use a smartphone device.
* Has access to a smartphone device running an operation system of Android 6 or above; or iOS 10 or above.

If taking part in the study through virtual visits, the following inclusion criteria also applies:

* Able to use, or has a caregiver who is able to use a personal computer, notebook or tablet.
* Has access to a personal computing device of that is:
* Running an operating system of macOS X with macOS 10.9 or later; or Windows 7 or above; or Ubuntu 12.04 or higher; or
* Have access to one of following internet browser software Internet Explorer version 11 or above; or Microsoft Edge version 12 or above; or Firefox version 27 or above; or Google Chrome version 30 or above; or Safari version 7 or above; capable of audio and video recording; and able to connect to the internet.

Exclusion Criteria:

* Clinically significant unstable psychiatric illness in 6 months.
* Diagnosis of General Anxiety Disorder.
* Current, or history within the past 2 years of major depressive disorder diagnosis (according to DSM-5 criteria); or psychiatric symptoms that, in the opinion of the investigator, could interfere with study procedures.
* History or presence of stroke within the past 2 years.
* Documented history of transient ischemic attack or unexplained loss of consciousness within the last 12 months.
* The participant is using drugs to treat symptoms related to AD, and the doses of these drugs were not stable for at least 8 weeks prior to consent.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified primarily through data-base searches of the Investigator sites.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the receiver operating characteristic (ROC) curve of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) Arms using speech recordings as input. | baseline

SECONDARY OUTCOMES:
The sensitivity of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) Arms. | baseline
The specificity of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) Arms. | baseline
The Cohen's kappa of the binary classifier distinguishing between amyloid positive (Arms 1 and 3) and amyloid negative (Arms 2 and 4) Arms. | baseline
The sensitivity of the binary classifier distinguishing between amyloid positive cognitively normal (CN) (Arm 3) and amyloid negative cognitively normal (CN) (Arm 4) Arms. | baseline
The specificity of the binary classifier distinguishing between amyloid positive cognitively normal (CN) (Arm 3) and amyloid negative cognitively normal (CN) (Arm 4) Arms. | baseline
The Cohen's kappa of the binary classifier distinguishing between amyloid positive cognitively normal (CN) (Arm 3) and amyloid negative cognitively normal (CN) (Arm 4) Arms. | baseline
The AUC of the binary classifier distinguishing between amyloid positive cognitively normal (CN) (Arm 3) and amyloid negative cognitively normal (CN) (Arm 4) Arms. | baseline
The sensitivity of the binary classifier distinguishing between amyloid positive MCI (Arm 1) and amyloid negative MCI (Arm 2) Arms. | baseline
The specificity of the binary classifier distinguishing between amyloid positive MCI (Arm 1) and amyloid negative MCI (Arm 2) Arms. | baseline
The Cohen's kappa of the binary classifier distinguishing between amyloid positive MCI (Arm 1) and amyloid negative MCI (Arm 2) Arms. | baseline
The AUC of the binary classifier distinguishing between amyloid positive MCI (Arm 1) and amyloid negative MCI (Arm 2) Arms. | baseline
The sensitivity of the binary classifier distinguishing between the MCI (Arms 1 and 2) and the CN (Arms 3 and 4) Arms. | baseline
The specificity of the binary classifier distinguishing between the MCI (Arms 1 and 2) and the CN (Arms 3 and 4) Arms. | baseline
The Cohen's kappa of the binary classifier distinguishing between the MCI (Arms 1 and 2) and the CN (Arms 3 and 4) Arms. | baseline
The AUC of the binary classifier distinguishing between the MCI (Arms 1 and 2) and the CN (Arms 3 and 4) Arms. | baseline
The agreement between the PACC5 composite and the corresponding regression model predicting it in all four Arms, as measured by the coefficient of individual agreement (CIA). | baseline
For each classifier/regressor in outcome 1-16, the correlation between the AUC/CIA and each age group, gender and speech-to-reverberation modulation energy ratio group, as measured by the Kendall rank correlation coefficient. | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emil Fristed, MSc, Principal Investigator — Novoic Limited
Locations (1):
- Syrentis Clinical Research, Santa Ana, California, United States

IPD SHARING:
Plan to Share IPD: Undecided